CLINICAL TRIAL: NCT00121017
Title: A Randomized, Open-Label Study Assessing Safety, Tolerability and Efficacy of an Induction-Maintenance Treatment Strategy Including Lopinavir/Ritonavir Plus Tenofovir Disoproxil Fumarate and Emtricitabine Versus Efavirenz Plus Tenofovir Disoproxil Fumarate and Emtricitabine in Antiviral-naïve HIV-1/HCV Co-Infected Subjects
Brief Title: A Study Exploring an Induction-Maintenance Kaletra-Based Therapy Versus a Sustiva-Based Regimen in Previously Non-Treated, HIV-1/HCV Co-Infected Subjects
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M05-731
Record Dates: First submitted 2005-07-14; First posted 2005-07-21 (Estimated); Last update posted 2006-07-27 (Estimated); Status verified 2006-07

CONDITIONS: HIV Infection; Hepatitis C
Keywords: HCV Infection; Treatment Naive
MeSH Terms: conditions — HIV Infections; Hepatitis C | interventions — lopinavir-ritonavir drug combination; Lopinavir; Ritonavir; efavirenz; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Tenofovir

INTERVENTIONS:
Drug: Kaletra (lopinavir/ritonavir)
Drug: Sustiva (efavirenz)
Drug: Truvada (emtricitabine/tenofovir disoproxil fumarate)

SUMMARY:
The purpose of this study is to determine whether a simplified lopinavir/ritonavir-based therapy will continue to keep the viral load at very low levels after initial treatment with a combination of Kaletra (lopinavir/ritonavir) plus tenofovir and emtricitabine.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age.
* Subject's plasma HIV-1 RNA is >1000 copies/mL at screening and in the investigator's opinion, the subject requires antiretroviral therapy.
* Subject is naive to antiretroviral therapy or has received <7 days total of any antiretroviral therapy >30 days prior to study drug administration.
* Subject has chronic HCV based on detectable plasma HCV RNA level (>600 IU/mL) at screening.
* Subject is not currently undergoing treatment of HCV infection and does not plan to initiate HCV treatment for the duration of this study.
* If female, the results of a urine pregnancy test performed at screening and on Day-1/Baseline are both negative.
* If female, subject is either not of childbearing potential, defined as postmenopausal for at least one year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or is of childbearing potential and practicing one of the following methods of birth control: condoms, sponge, foams, jellies, diaphragm or intrauterine device, a vasectomized partner or total abstinence from sexual intercourse.
* Subject is not breastfeeding.
* Subject's vital signs, physical examination and laboratory results do not exhibit evidence of acute illness.
* Subject agrees not to take any drugs during the study, including over-the-counter medicines, vitamins, mineral supplements, herbal preparations, alcohol or recreational drugs without the knowledge and permission of the investigator.
* Subject has not been treated for an active AIDS-defining opportunistic infection within 30 days of initiating study drug.
* Subject has voluntarily signed and dated an informed consent from, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), after the nature of the study has been explained and the subject has had the opportunity to ask questions. The informed consent must be signed before any study-specific procedures are performed.

Exclusion Criteria:

* Subject has a history of an allergic reaction or significant sensitivity to lopinavir, ritonavir, tenofovir, emtricitabine, lamivudine, and efavirenz or to any inert materials contained in the study drug formulations.
* Subject has a significant history of cardiac, renal, neurologic, psychiatric, oncologic or metabolic disease that would, in the opinion of the investigator, adversely affect his/her participation in this study.
* Subject has chronic hepatic disease of any etiology other than HCV infection (including hemochromatosis, autoimmune hepatitis, Wilson's Disease, and hepatocellular carcinoma).
* Subject has a liver biopsy result consistent with advanced chronic cirrhosis or a Child Pugh Score of "C".
* Subject is currently taking or will require any drugs that are contraindicated or have significant pharmacokinetic interactions with study drugs during the course of the study. For complete information refer to the most current product label for locally approved prescribing information for lopinavir/ritonavir (Kaletra), efavirenz (Sustiva), tenofovir disoproxil fumarate (Viread), emtricitabine (Emtriva), co-formulated emtricitabine/tenofovir disoproxil fumarate (Truvada) and lamivudine (Epivir).
* Subject has ongoing history of drug and/or alcohol abuse or psychiatric illness that in the investigator's opinion could preclude compliance with the protocol.
* Subject has received any investigational drug or vaccine within 30 days prior to study drug administration.
* The screening HIV-1 genotype resistance report suggests resistance or possible resistance to the study RTI(s) or lopinavir/ritonavir; Evidence of possible resistance to efavirenz; Presence of one of the following mutations: RT L1001, K103N, V106A or M, V108I, Y181C or I, Y188L, G190A or S, P225H, M230L; Evidence of possible resistance to emtricitabine or lamivudine; Presence of one of the following mutations: RTm184V or I; Evidence of possible resistance to tenofovir; Presence of RT K65R or insertion at codon 69, or Presence of 2 or more of the following mutations: RTm41L, D67N, K70R, L210W; any change at T215, K219Q or evidence of possible resistance to lopinavir/ritonavir; Presence of one or more of the following mutations: protease I47V or A, G48V, I50V, V82A or F or T or S, I84V, 190M or Presence of 3 or more of the following mutations: protease L10F or I or R or V, K20M or R, L24I, V32I, L33F, M36I, M46I or L, F53L; any change at I54, A71V or T, G73S.
* Screening laboratory analyses show any of the following abnormal laboratory results: Presence of hepatitis B surface antigen (HBsAg) or anti-HBcAB (Total Ig, Total Bilirubin >/= 2.5x upper limit of normal (ULN), Hemoglobin <8.0 g/dL, Absolute neutrophil count < 750 cells/uL, Platelet count < 50,000/mL, ALT (SGPT) or AST (SGOT) > 5.0x ULN, Creatinine > 1.5x ULN, Calculated creatinine clearance < 50 mL/min, PT > 3.0 seconds prolonged from the ULN.
* For any reason, subject is considered by the investigator to be an unsuitable candidate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200

PRIMARY OUTCOMES:
The proportion of subjects with a plasma HIV-1 RNA level below 50 copies/mL at Week 96.

SECONDARY OUTCOMES:
Vital signs
Physical examinations
Clinical laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information, Study Director — Abbott